CLINICAL TRIAL: NCT03262220
Title: Pilot Study of Dose Escalated Total Marrow Irradiation With Volumetric Arc Therapy for Patients With Hematological Malignancies Unfit for a Standard 12 Gy TBI Conditioning Regimen.
Brief Title: Total Marrow Irradiation With Volumetric Arc Therapy for Patients Unfit for a 12 Gy TBI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Thomas Zilli (Other)
Collaborators: University Hospital, Geneva (Other)
Responsible Party: Sponsor-Investigator, Thomas Zilli, MD, PD, Médecin Adjoint Agrégé, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-00066
Record Dates: First submitted 2017-08-23; First posted 2017-08-25 (Actual); Last update posted 2020-05-14 (Actual); Status verified 2020-05

CONDITIONS: Haematological Malignancy
Keywords: Haematological malignancy; Total Marrow Irradiation; Volumetric Arc Therapy
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: Volumetric Arc Therapy (VMAT) — Total Marrow Irradiation: 12 Gy in 3 fractions of 4 Gy on 3 consecutive days with a concomitant simultaneous integrated boost (SIB) of 4.5 Gy x 3 fractions delivered to active bone marrow (ABM).

SUMMARY:
Total body irradiation (TBI) is a standard part of the conditioning regimen for bone marrow transplantation (BMT). Several randomized trials have shown superior outcomes using TBI compared with non TBI-containing regimens. Standard TBI is usually delivered over three days for a total dose of 12 Gy with two daily fractions. However, as demonstrated by our group, increasing the TBI dose above 10 Gy is not necessarily associated with better outcome in patients undergoing allogenic BMT for hematologic malignancies. For this reason, patients older than 40 or grafted after relapse are treated at our center with a reduced-dose 10 Gy TBI regimen. This pilot study wishes to investigate in 10 patients with hematological malignancies unfit for a standard 12 Gy TBI conditioning regimen a more targeted, conformal form of treatment, referred as total marrow (TMI), using volumetric Arc Therapy (VMAT). Our hypothesis is that using this technique that can allow deliver a higher total dose to the target while at the same time assuring to the organs at risk (OAR) the same dose normally delivered with a 10 Gy TBI we will improve the therapeutic ratio in these patients.

DETAILED DESCRIPTION:
This is a feasibility prospective pilot study. Ten patients ≥ 40 years with hematologic malignancies prior to Bone Marrow Transplant (BMT) will receive a dose escalated hypofractionated Total Marrow Irradiation (TMI) (12 Gy in 3 fractions, daily, on 3 consecutive days).

The current project is a joint initiative in translational and clinical medical research between the Radiation-oncology workgroup and the Bone Marrow transplant workgroup of University Hospitals of Geneva (HUG).

ELIGIBILITY:
Inclusion Criteria:

* Karnofsky performance status ≥ 70
* Presence of any kind of haematological malignancy in complete remission (CR1, CR2 ore CR3) at time of transplantation, with the exception of patients with myelodysplastic syndrome.
* Patients that are scheduled for a BMT either using stem cell derived from bone marrow or peripheral blood stem cells.
* Candidates to receive a 10 Gy TBI treatment.
* Ability to stay still and lying on the treatment couch for at least 45 minutes.
* Informed Consent as documented by signature.

Exclusion Criteria:

* Karnofsky performance status <70 intended as a patient unable to work; able to live at home and care for most personal needs with varying amount of assistance needed.
* Concurrent treatment with other experimental drugs or other anti-cancer therapy.
* Participation in another clinical trial and any concurrent treatment with any investigational drug within 4 weeks prior to trial entry/randomisation.
* Inability to comply with study and follow-up procedures.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2017-04-11 (Actual); Primary Completion 2021-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Grade II and III toxicity | 30 days after radiotherapy
  (Seattle Regimen-related toxicity grade) 30 days after transplant in patients with hematologic malignancies treated with a dose-escalated hypofractionated VMAT-based TMI

SECONDARY OUTCOMES:
Cumulative incidence of Transplant Related Mortality(TRM) | 100 days post-bone marrow transplantation
  Defined as death occurring from causes that are different other than disease relapse post-transplant
Cumulative incidence of Grade II Organ toxicity | up to day 100 post-bone marrow transplantation
  Seattle Regimen-related toxicity grade

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Geneva, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No
No plan